CLINICAL TRIAL: NCT04573075
Title: Is a Ghost Ileostomy a Safe Alternative to a Protective Loop Ileostomy for Patients After Colorectal Resections ?
Brief Title: Ghost Ileostomy (GI) Versus Loop Ileostomy (LI) After Colorectal Resections
Acronym: GI_versus_LI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelisches Klinikum Köln Weyertal gGmbH (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Principal Investigator, Claudia Rudroff, Head of the Department for Visceral Surgery and Surgery of the lower Gastrointestinal Tract, Evangelisches Klinikum Köln Weyertal gGmbH
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI_observational_01_20
Record Dates: First submitted 2020-09-12; First posted 2020-10-05 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Surgery
Keywords: ghost ileostomy; loop ileostomy; colorectal resection
MeSH Terms: interventions — Ileostomy

STUDY DESIGN:
Intervention Model Description: Ghost ileostomy (short: ghost stoma) as an alternative to protective loop ileostomy or no outlet after colorectal resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no outlet (Other): no outlet is used after colorectal resection and forming of a primary anastomosis
  Interventions: Procedure: no outlet
- loop ileostomy (Active Comparator): loop ileostomy is applied after colorectal resection and forming of a primary anastomosis
  Interventions: Procedure: loop ileostomy
- ghost ileostomy (Experimental): ghost ileostomy or ghost stoma (synonyms) is performed after colorectal resection and forming of a primary anastomosis
  Interventions: Procedure: Ghost ileostomy

INTERVENTIONS:
Procedure: Ghost ileostomy — a loop of the small bowel is marked with a silicone strap and externalized through the abdominal wall to avoid a loop ileostomy
  Other Names: Ghost stoma
  Arms: ghost ileostomy
Procedure: loop ileostomy — a protective loop ileostomy is applied after after colorectal resection and forming of a primary anastomosis
  Arms: loop ileostomy
Procedure: no outlet — no further intervention is used after colorectal resection and forming of a primary anastomosis
  Arms: no outlet

SUMMARY:
A Ghost Ileostomy (GI) as an alternative to a diverting protective Loop Ileostomy (LI) after colorectal resection is offered the patients at risk preoperatively. A GI is only applied in cases, who would receive a LI otherwise.

DETAILED DESCRIPTION:
A protective loop ileostomy (LI) is applied to protect a critical anastomosis after left sided colorectal resections. It is routinely indicated after low anterior rectal resection because this location carries a high risk for anastomotic insufficiency due to poor blood supply and tension of the bowel itself. A LI is also used to protect a primary anastomosis after other colorectal resections, if the surgeon in charge deems it necessary. However, the LI does not reduce the rate of insufficiencies (between 8-18%), but decreases the rate and severity of the associated complications and its mortality.

Furthermore, the LI is associated with complications of its own. Stoma malfunction due to torsion may cause a bowel obstruction, local complications may lead to an abscess or wound dehiscence, and in the long term follow-up surgical interventions due to hernias at the stoma site or adhesions with a consecutive ileus may become necessary.

Additionally, many patients are traumatized by the thought of a stoma. Thus, the routine application of a LI is currently critically discussed and its need re-evaluated.

A Ghost ileostomy (GI) is an alternative. Instead of a real diverting stoma the suitable small bowel loop is marked with a silicon strap, which is externalized through the abdominal wall and fixed with sutures. No real stoma outlet needs to be formed. In case of an anastomotic leakage (AL) the GI is easily converted to a LI by extracting the marked bowel loop through the abdominal wall. Besides increasing patients' comfort, ileostomy-related morbidity, hospital re-admissions for the closure of the ileostomy, and health care expenses related to the stoma supply and complications can be avoided.

In a recent systematic review of the existing literature Baloyiannis et al. identified 11 studies with altogether 554 patients. They found a total complication rate of 13.9%, with 2,1% GI-specific adverse events. Although it is a safe and comfortable option for low- and medium-risk patients it is still not established routinely.

Aim of the study:

The study wants to examen whether the routine use of a GI after colorectal resection with primary anastomosis can reduce the number of LI needed. This should avoid the stoma associated complications and the re-hospitalization for the stoma closure. A further endpoint is the routine use of GI as an alternative has to ensure patients safety. No further risk should result from this new intervention.

Study design:

Prospective clinical observational study

Method:

All patients after a colorectal resection with a primary anastomosis are offered the option of a GI as an alternative to a LI preoperatively. They have to consent in a stoma, if the surgeon in charge deems this necessary during the procedure. Written informed consent is obtained prior to surgery. At the end of the colorectal resection the surgeon in charge decided whether to shape a GI, a LI or no outlet. General criteria for a stoma are a redo anastomosis, an ultralow rectal resection, peritonitis at the site of the anastomosis, or an extended endometriosis resection in the pelvis. In case of emergency surgery a Hartman procedure may become necessary due to the critical condition of the patient. A GI is only applied in cases, who would have received a LI otherwise.

Technically, a silicon loop (Roeser Loops super maxi, Ref No 10.11522; Roeser Medical GmbH, Bochum, Germany; conformity european (CE) 0481) marks a suitable terminal ileum loop and is externalized through the 5 m trocar site regularly placed in the right upper quadrant of the abdomen or a similar mini-incision in cases of open surgery. The loop is fixed with two penetrating, non-absorbable sutures and closed with a wound dressing.

Postoperatively patients are observed on the intensive care unit (ICU) for 12-48 hours. Further action - ultrasound, CT scan, and/or colonoscopy - is taken in cases of fever, laboratory signs of inflammation (leucocyte count >15x1000ul, procalcitonin >1 ng/ml, or C-reactive protein more than three times the initial value). Pelvic fluid collection, bowel malfunction, or signs of anastomotic leakage will lead to a re-operation converting the GI to a LI and an abdominal lavage with drainage, if necessary. In all other cases of GI the silicon strap will be removed after the initiation of bowel function.

All patients included will be asked about their well being and medical treatments related to their colorectal resection after their dismission in a follow-up phone call 6 months after surgery. The study ends with this last survey.

ELIGIBILITY:
Inclusion Criteria:

* informed consent

Exclusion Criteria:

* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participants eligibility is based in self-representation of gender identity
Enrollment: 257 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
number of protective loop ileostomies avoided by the ghost stoma | through study completion, an average of one year
  The number of ghost ileostomies that did not need to be transformed to a loop ileostomy is counted.

SECONDARY OUTCOMES:
Morbidity and Mortality after ghost ileostomy compared to the other groups | through study completion, an average of one year
  Surgical outcome measured concerning the postoperative morbidity and mortality according to the Clavien Dindo classification (CDC). CDC distinguishes: no complication = 0; mild complication without further intervention needed = 1; mild complication with medication like antibiotics needed=2; complication with further intervention needed =3a, complication with further intervention under general anesthesia needed =3b; septic complication =4; death =5.

OTHER OUTCOMES:
health care expenses | through study completion, an average of one year
  the amount of health care expenses spared by applying a ghost stoma compared to the general costs of a stoma closure, if applicable; results are expressed in €s per case
participants' satisfaction with the experimental intervention | through study completion, an average of one year
  measurement of participants satisfaction on a scale between 1 (not satisfied at all) to 4 (very satisfied)
operating time needed in cases of a ghost ileostomy | through study completion, an average of one year
  operating time in minutes of the group with a GI compared to the group with an LI and the group with no outlet

CONTACTS AND LOCATIONS:
Overall Officials: Claudia L Rudroff, PhD MD, Principal Investigator — EVK Koeln
Locations (1):
- Evangelisches Klinikum Koeln Weyertal, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDermott FD, Heeney A, Kelly ME, Steele RJ, Carlson GL, Winter DC. Systematic review of preoperative, intraoperative and postoperative risk factors for colorectal anastomotic leaks. Br J Surg. 2015 Apr;102(5):462-79. doi: 10.1002/bjs.9697. Epub 2015 Feb 19. PMID 25703524
- [Background] Ihnat P, Gunkova P, Peteja M, Vavra P, Pelikan A, Zonca P. Diverting ileostomy in laparoscopic rectal cancer surgery: high price of protection. Surg Endosc. 2016 Nov;30(11):4809-4816. doi: 10.1007/s00464-016-4811-3. Epub 2016 Feb 22. PMID 26902615
- [Background] Sacchi M, Legge PD, Picozzi P, Papa F, Giovanni CL, Greco L. Virtual ileostomy following TME and primary sphincter-saving reconstruction for rectal cancer. Hepatogastroenterology. 2007 Sep;54(78):1676-8. PMID 18019692
- [Result] Hernandez AV, Otten J, Christ H, Ulrici C, Piriyev E, Ludwig S, Rudroff C. Ghost Ileostomy: Safe and Cost-effective Alternative to Ileostomy After Rectal Resection for Deep Infiltrating Endometriosis. In Vivo. 2022 May-Jun;36(3):1290-1296. doi: 10.21873/invivo.12829. PMID 35478159
- See also: Standard operating procedure on the treatment of colorectal cancer in Germany — https://www.awmf.org/leitlinien/detail/ll/021-007OL.html